CLINICAL TRIAL: NCT02165267
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Drug Levels of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01) Administered in Multiple Doses Intravenously and Subcutaneously in Different Dosing Schedules to Healthy, HIV-Uninfected Adults
Brief Title: Evaluating the Safety and Drug Levels of an Antibody Against HIV in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 104; 11969 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1: VRC01 (6 IV infusions) (Experimental): Participants will receive an IV infusion of 40 mg/kg of VRC01 administered in 100 mL of normal saline over 1 hour at Day 0, followed by IV infusions of 20 mg/kg of VRC01 administered in 100 mL of normal saline over at least 30 minutes to 1 hour at Days 28, 56, 84, 112, and 140.
  Interventions: Biological: VRC01
- Arm 2: VRC01 (3 IV infusions) (Experimental): Participants will receive an IV infusion of 40 mg/kg of VRC01 administered in 100 mL of normal saline over 1 hour at Day 0 and over at least 30 minutes to 1 hour at Days 56 and 112.
  Interventions: Biological: VRC01
- Arm 3a: VRC01 (1 IV infusion plus multiple SC injections) (Experimental): Participants will receive an IV infusion of 40 mg/kg of VRC01 administered in 100 mL of normal saline over 1 hour at Week 0, followed by SC injection of 5 mg/kg of VRC01 administered every 2 weeks for 20 weeks.
  Interventions: Biological: VRC01
- Arm 3b: Placebo for VRC01 (infusion plus injections) (Placebo Comparator): Participants will receive an IV infusion of sodium chloride placebo administered in 100 mL of normal saline over 1 hour at Week 0, followed by SC injection of placebo for VRC01 administered every 2 weeks for 20 weeks.
  Interventions: Biological: SC placebo for VRC01; Biological: IV placebo for VRC01
- Arm 4: 10 mg/kg of VRC01 (3 IV infusions) (Experimental): Participants will receive an IV infusion of 10 mg/kg of VRC01 administered in 100 mL of normal saline over 1 hour at Month 0 and over at least 30 minutes to 1 hour at Months 2 and 4.
  Interventions: Biological: VRC01
- Arm 5: 30 mg/kg of VRC01 (3 IV infusions) (Experimental): Participants will receive an IV infusion of 30 mg/kg of VRC01 administered in 100 mL of normal saline over 1 hour at Month 0 and over at least 30 minutes to 1 hour at Months 2 and 4.
  Interventions: Biological: VRC01

INTERVENTIONS:
Biological: VRC01 — Administered IV in 100 mL of normal saline (Sodium Chloride for Injection 0.9%, USP) or administered SC by needle and syringe injection.
  Other Names: Human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB
  Arms: Arm 1: VRC01 (6 IV infusions); Arm 2: VRC01 (3 IV infusions); Arm 3a: VRC01 (1 IV infusion plus multiple SC injections); Arm 4: 10 mg/kg of VRC01 (3 IV infusions); Arm 5: 30 mg/kg of VRC01 (3 IV infusions)
Biological: SC placebo for VRC01 — Sterile, buffered aqueous solution of 25 mM Sodium Citrate, 50 mM Sodium Chloride, 150 mM L-Arginine Hydrochloride, 10% Dextran 40, and 0.005% Polysorbate 80 at pH 5.8 administered SC by needle and syringe injection
  Other Names: SC placebo for VRC-PLAMAB068-00-AB
  Arms: Arm 3b: Placebo for VRC01 (infusion plus injections)
Biological: IV placebo for VRC01 — Sodium Chloride for Injection 0.9%, USP administered IV in 100 mL of normal saline (Sodium Chloride for Injection 0.9%, USP)
  Other Names: Sodium Chloride for Injection 0.9%, USP
  Arms: Arm 3b: Placebo for VRC01 (infusion plus injections)

SUMMARY:
Antibodies are natural proteins that the body makes to fight infections. Antibodies can also be manufactured like a drug and infused or injected into the body to prevent or treat a disease. The purpose of this study is to test the safety of and the body's response to an antibody against HIV in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and drug levels of five different schedules for the intravenous (IV) and subcutaneous (SC) administration of a human monoclonal antibody (VRC-HIVMAB060-00-AB [VRC01]) against HIV in healthy, HIV-uninfected adults.

The study will enroll 88 healthy, HIV-uninfected adults aged 18 to 50 years.

This study will enroll participants in 5 groups. Groups 1-3 will enroll simultaneously. Groups 1 and 2 will be randomized together but not blinded, while Group 3 will be randomized separately and will be blinded. With the implementation of Version 2.0, Groups 4 and 5 will be randomized together and will enroll simultaneously. Each group will have a different schedule of clinic visits and receive different doses of VRC01 or placebo for VRC01. Participants will attend 8 months of scheduled clinic visits.

Participants in Group 1 will receive an IV infusion of VRC01 on Days 0, 28, 56, 84, 112, and 140. Participants in Group 2 will receive an IV infusion of VRC01 on Days 0, 56, and 112. Participants in Group 3 will receive an IV infusion of VRC01 or IV placebo for VRC01 on Day 0, followed by SC injections of VRC01 or SC placebo for VRC01 on Days 14, 28, 42, 56, 70, 84, 98, 112, 126, 140, and 154. Participants in Groups 4 and 5 will receive an IV infusion of VRC01 (each group will receive a different dose) on Days 0, 56, and 112.

Participants will remain in the clinic for about an hour after receiving the infusions and injections for observation and monitoring. Participants in Group 3 who have no problems with the first SC injection will have to wait in the clinic for only a half an hour after the rest of the SC injections.

At study entry, participants will give a medical history; undergo a physical exam, blood collection, and urine collection; and receive HIV risk reduction counseling. At follow-up visits, participants will undergo a brief physical exam and blood collection, receive HIV risk reduction counseling, and be asked questions about their health and their experience participating in the study. At all visits, participants who were born female will have a pregnancy test. At select study visits, saliva, rectal, and semen or cervical secretion samples will be collected from participants who consent to collection of these samples.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Weight at least 53 kg and up to 115 kg
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first infusion, with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until completion of the last study visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit

Laboratory Inclusion Values

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female, greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell count equal to 2,500 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to the institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: U.S. participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus (anti-HCV) antibodies, or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cell levels within institutional normal range).

Reproductive Status

* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (beta-HCG) pregnancy test performed prior to infusion on the day of initial infusion. Persons who are not of reproductive potential because of having undergone total hysterectomy with bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
* Reproductive status: A participant who was born female must:

  * Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using any of the following methods: condoms (male or female) with or without a spermicide; diaphragm or cervical cap with spermicide; intrauterine device (IUD); hormonal contraception; any other contraceptive method approved by the HVTN 104 Protocol Safety Review Team (PSRT); successful vasectomy in the male partner (considered successful if a participant reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit.

Exclusion Criteria:

General

* Blood products received within 120 days before first infusion, unless eligibility for earlier enrollment is determined by the HVTN 104 PSRT
* Investigational research agents received within 30 days before first infusion
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 104 study
* Pregnant or breastfeeding

Vaccines and Other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 104 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 6 months in a prior vaccine trial. Exceptions may be made for some vaccines and vaccine trials. For participants who have received an experimental vaccine(s) less than 6 months ago, eligibility for enrollment will be determined by the HVTN 104 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 10 days before first infusion and with no evidence of residual inflammation; or scheduled within 10 days after first infusion (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever).
* Previous receipt of humanized or human monoclonal antibodies (mAbs) whether licensed or investigational

Immune System

* Immunosuppressive medications received within 30 days before first infusion. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days, with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines or to vaccine components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child)
* Immunoglobulin received within 90 days before first infusion, unless eligibility for earlier enrollment is determined by the HVTN 104 PSRT.
* Autoimmune disease (Not excluded: participant with mild, stable, and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate reactogenicity and adverse event [AE] assessments)
* Immunodeficiency

Clinically Significant Medical Conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated infusions or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma (symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program [NAEPP] Expert Panel report).
* Exclude a participant who uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or uses moderate/high dose inhaled corticosteroids, or in the past year has either of the following:

  * Greater than one exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: history of seizure(s) within past 3 years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Assessment of local and systemic reactogenicity signs and symptoms | Measured through Month 5.5 visit
  Assessment occurs at each product administration and for 3 days after administration.
Measurements of laboratory measures of safety | Measured through participants' last study visit at Month 8
Assessment of adverse events | Measured through participants' last study visit at Month 8
Assessment of serious adverse events | Measured through participants' last study visit at Month 8
Number of early discontinuation of infusions | Measured through participants' last study visit at Month 8
  The assessment will include the reason(s) for discontinuation of infusions and early study termination.
Serum concentration of VRC01 in Groups 1-3 at Month 6 | Measured at Month 6
Serum concentration of VRC01 28 and 56 days after each IV administration in Groups 4 and 5 | Measured 56 days after each IV administration

SECONDARY OUTCOMES:
Magnitude of serum neutralization of a single VRC01 sensitive virus isolate as measured in the TZMbl assay at multiple timepoints | Measured through participants' last study visit at Month 8
Serum concentration of VRC01 in each group at multiple timepoints | Measured through participants' last study visit at Month 8
Serum concentration of anti-VRC01 antibodies in each group at multiple timepoints compared to corresponding VRC01 levels | Measured through participants' last study visit at Month 8
Mucosal levels of VRC01 in each group at multiple timepoints | Measured through participants' last study visit at Month 8
Magnitude of neutralization in genital, rectal, and oral secretions of a single VRC01 sensitive virus isolate as measured in the TZMbl assay at multiple timepoints | Measured through participants' last study visit at Month 8
Assessment of VRC01 binding in serum and genital, rectal, and oral secretions to multiple Env proteins in each group at multiple timepoints (assessed by binding antibody multiplex assay) | Measured through participants' last study visit at Month 8

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mayer, Study Chair — The Fenway Institute
Locations (6):
- United States (6):
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Mayer KH, Seaton KE, Huang Y, Grunenberg N, Isaacs A, Allen M, Ledgerwood JE, Frank I, Sobieszczyk ME, Baden LR, Rodriguez B, Van Tieu H, Tomaras GD, Deal A, Goodman D, Bailer RT, Ferrari G, Jensen R, Hural J, Graham BS, Mascola JR, Corey L, Montefiori DC; HVTN 104 Protocol Team; and the NIAID HIV Vaccine Trials Network. Safety, pharmacokinetics, and immunological activities of multiple intravenous or subcutaneous doses of an anti-HIV monoclonal antibody, VRC01, administered to HIV-uninfected adults: Results of a phase 1 randomized trial. PLoS Med. 2017 Nov 14;14(11):e1002435. doi: 10.1371/journal.pmed.1002435. eCollection 2017 Nov. PMID 29136037